CLINICAL TRIAL: NCT05720754
Title: Safety and Efficacy of Heated Artificial Tears Under Practical Conditions
Brief Title: Temperature on Evaporative Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDEDQS2023
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye
Keywords: dry eye; heated eye mask; diquafosol; tear breakup time; ocular surface disease index
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Masked examiner for all clinical assessments will not involved in the data collection or group allocation procedure for this research. The investigator will not be aware of the three groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DQS+HEM (Experimental): Participants in the DQS+ group used DQS 1 drop 3 times/per day with heated eye mask for 2 weeks
  Interventions: Drug: Diquafosol tetrasodium; Device: Heated eye mask
- DQS (Active Comparator): Participants in the DQS group used DQS 1 drop 3 times/per day for 2 weeks
  Interventions: Drug: Diquafosol tetrasodium
- HEM (Active Comparator): Participants in the HEM group used heated eye mask 3 times/per day for 2 weeks
  Interventions: Device: Heated eye mask

INTERVENTIONS:
Drug: Diquafosol tetrasodium — 3% Diquafosol tetrasodium eye drops will be used to assess its usefulness in dry eye signs and symptoms
  Other Names: Diquas
  Arms: DQS; DQS+HEM
Device: Heated eye mask — Heated eye mask will be used to assess its usefulness in dry eye signs and symptoms
  Arms: DQS+HEM; HEM

SUMMARY:
Ocular surface temperature of a normal person is around 34.6 degree centigrade. After instilling the eye drop, depending on the temperature of the eye drop and the ocular surface, the ocular surface temperature will temporally increase or decrease sightly. Warm feeling will make blood vessels dilated and more blood will pass through to bring more blood flow out of our body to the heated area of the body and makes cells more permeable. Therefore, heating the ocular surface with heated eye mask after instilling artificial tears has the possibility to improve drug permeability on the ocular surface.

DETAILED DESCRIPTION:
Evaporative dry eye (EDE) is common and can lead to ocular pain, decreased visual quality, and reduced quality of life. 3% diquafosol (DQS) ophthalmic solution and heated eye mask (HEM) have been found to be beneficial in reducing signs and symptoms of dry eye. Warm compress therapy temperature of 40 °C to 45 °C have been typically advocated to melt the meibium causing obstruction at the orifices of the meibomian gland, eventually allowing increased lipid layer of the tear film. While in impact of heat on the ocular surface (OS) has not been extensively studied. Controlled and precise application of heat has the ability to create a cascade of events in the skin and thus aids in facilitating a faster movement of molecules into and across the skin. Possible mechanisms of enhancing drug permeation include on the ocular surface could be: (mechanisms may operate individually or concurrently):

* increase in drug diffusivity in the vehicle and/or in the ocular surface
* increase in partitioning and diffusion
* alteration in the lipid structure
* increased local blood flow Therefore, the purpose of this RCT is to assess the impact of instilling 3% DQS ophthalmic solution follow by HEM raising the OS temperature by 40 degrees centigrade for 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* The presence of at most one symptom including burning, foreign body sensation, itching or eye fatigue for 3 months
* OSDI score ≥ 13 and TBUT <5 s or NIBUT < 10s
* Able and willing to comply with the treatment/follow-up schedule

Exclusion Criteria:

* A recent history (past 30 days) of topical ophthalmic medication use, including antibiotics, steroids, non-steroidal anti-inflammatory drugs, or required the chronic use of topical ophthalmic medications
* Eyelids or intraocular tumors that should not put pressure
* Active allergy or infection or inflammatory disease that may have prevented the subjects from completing the study at the ocular surface
* Any structural change in lacrimal passage
* Glaucoma
* Diabetes or other systemic, dermatologic, or neurologic diseases that affect the health of ocular surface
* Use of any systemic anti-inflammatory drugs or medication that may interfere with tear production, such as antianxiety, antidepressive, and antihistamine medications within 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-04-02 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Non-invasive tear break-up time (NIBUT) | Day-0 (baseline), day-7, and day-14
  Non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Ocular Surface Disease Index (OSDI) | Day-0 (baseline), day-7, and day-14
  OSDI, which is a questionnaire consisting of 12 questions for evaluating the effects of dry eye syndrome on vision, ocular symptoms and any condition associated with DED. The patient will answer each question on a scale ranging from 0 to 4, with 0 indicating 'none of the time' and 4 indicating 'all of the time'. If a certain question is deemed irrelevant, it will be marked as 'not applicable (N/A)' and excluded from the analysis. The OSDI total score is calculated according to the following formula. The scale ranges from 0 to 100, with higher scores representing more severe cases of dry eye syndrome.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined

SECONDARY OUTCOMES:
Fluorescein and lissamine conjunctival and cornea staining (CFS) | Day-0 (baseline), day-7, and day-14
  Fluorescein and lissamine staining of the ocular surface will be divided into three zones comprising nasal conjunctival, corneal, and temporal conjunctival areas. The staining score ranged from 0 to 3 for each zone, yielding a total score of 0-9 for the ocular surface.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Meibomian gland function and secretion quality | Day-0 (baseline), day-7, and day-14
  Meibum quality will be assessed under a slit-lamp: Five meibomian gland in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste like consistency meibum)
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Tear Film Lipid Layer Score (TFLL) | Day-0 (baseline), day-7, and day-14
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan). The results will be graded as follows: grade 1, somewhat gray color, uniform distribution; grade 2, somewhat gray color, nonuniform distribution; grade 3, a few colors, nonuniform distribution; grade 4, many colors, nonuniform distribution; grade 5, corneal surface partially exposed.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Tear meniscus height (TMH) | Day-0 (baseline), day-7, and day-14
  Non-invasive first tear film breakup time using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively and the median value was recorded.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Conjunctival hyperemia (RS score) | Day-0 (baseline), day-7, and day-14
  Conjunctival hyperemia (RS score) will be assessed by Keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 (normal) to 4.0 (severe).
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Eric Pazo, MD, PhD, Study Chair — He Eye Hospital, Shenyang, China
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
The study's findings will be shared regardless of the effect's direction. All possible beneficiaries of the research, including patients, carers, family, doctors, advisory boards, and medical boards, will receive trial data. Publications in high impact, open-access medical journals and talks at national and international medical conferences will serve this purpose.
Supporting Information: Study Protocol, SAP
Time Frame: The Steering Committee will write and submit the report for publication at the end of the study
Access Criteria: Use in clinical studies

REFERENCES:
- [Result] Ma J, Pazo EE, Zou Z, Jin F. Prevalence of symptomatic dry eye in breast cancer patients undergoing systemic adjuvant treatment: A cross-sectional study. Breast. 2020 Oct;53:164-171. doi: 10.1016/j.breast.2020.07.009. Epub 2020 Aug 5. PMID 32836200
- [Result] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Result] Bron AJ, Tiffany JM. The contribution of meibomian disease to dry eye. Ocul Surf. 2004 Apr;2(2):149-65. doi: 10.1016/s1542-0124(12)70150-7. PMID 17216085
- [Result] Chhadva P, Goldhardt R, Galor A. Meibomian Gland Disease: The Role of Gland Dysfunction in Dry Eye Disease. Ophthalmology. 2017 Nov;124(11S):S20-S26. doi: 10.1016/j.ophtha.2017.05.031. PMID 29055358
- [Result] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Result] Kulkarni AA, Trousdale MD, Stevenson D, Gukasyan HJ, Shiue MH, Kim KJ, Read RW, Lee VH. Nucleotide-induced restoration of conjunctival chloride and fluid secretion in adenovirus type 5-infected pigmented rabbit eyes. J Pharmacol Exp Ther. 2003 Jun;305(3):1206-11. doi: 10.1124/jpet.103.049221. Epub 2003 Mar 20. PMID 12649304
- [Result] Dota A, Sakamoto A, Nagano T, Murakami T, Matsugi T. Effect of Diquafosol Ophthalmic Solution on Airflow-Induced Ocular Surface Disorder in Diabetic Rats. Clin Ophthalmol. 2020 Apr 1;14:1019-1024. doi: 10.2147/OPTH.S242764. eCollection 2020. PMID 32280196
- [Result] Jumblatt JE, Jumblatt MM. Regulation of ocular mucin secretion by P2Y2 nucleotide receptors in rabbit and human conjunctiva. Exp Eye Res. 1998 Sep;67(3):341-6. doi: 10.1006/exer.1998.0520. PMID 9778415
- [Result] Tanioka H, Kuriki Y, Sakamoto A, Katsuta O, Kawazu K, Nakamura M. Expression of the P2Y(2) receptor on the rat ocular surface during a 1-year rearing period. Jpn J Ophthalmol. 2014 Nov;58(6):515-21. doi: 10.1007/s10384-014-0342-4. Epub 2014 Sep 2. PMID 25179431
- [Result] Cowlen MS, Zhang VZ, Warnock L, Moyer CF, Peterson WM, Yerxa BR. Localization of ocular P2Y2 receptor gene expression by in situ hybridization. Exp Eye Res. 2003 Jul;77(1):77-84. doi: 10.1016/s0014-4835(03)00068-x. PMID 12823990